CLINICAL TRIAL: NCT05159778
Title: A Multicenter, Open-label, Phase 2 Study of Imprime PGG and Pembrolizumab in Patients With Metastatic Breast Cancer (mBCA) Who Have Progressed Through Prior Hormonal Therapy
Brief Title: Phase 2 Study of Imprime PGG and Pembrolizumab in Patients With HR+/HER2- Metastatic Breast Cancer (mBCA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGG-BCA2121 / MK-3475-C99
Record Dates: First submitted 2021-11-10; First posted 2021-12-16 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-07

CONDITIONS: Malignant Neoplasm of Breast
Keywords: ER/PR+/ HER2(-) metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — BTH1677; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open label Simon 2 stage design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Biological: Imprime PGG; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Imprime PGG — Imprime PGG is a soluble, β-1,3/1,6 glucan isolated from the cell wall of a proprietary Saccharomyces cerevisiae yeast strain. Imprime PGG acts as a Pathogen-Associated Molecular Pattern (PAMP). Imprime will be administered at a dose of 4 mg/kg IV over a 2-hour infusion time on Days 1, 8 and 15 of each 3-week treatment cycle.
  Other Names: Imprime; BTH-1677
Biological: Pembrolizumab — Pembrolizumab is a humanized monoclonal antibody against the programmed death receptor-1 protein. Pembrolizumab will be given at a fixed dose of 200 mg IV over 30 minutes on Day 1 of each 3-week treatment cycle after the Imprime infusion.
  Other Names: Keytruda

SUMMARY:
The primary objective of this Phase 2 Simon 2-Stage study is to determinate the Overall Response Rate (ORR) per RECIST v1.1 following treatment with Imprime PGG + pembrolizumab in patients with ER/PR+/ HER2(-) metastatic breast cancer who have progressed through prior hormone therapy with at least one CDK4/6 inhibitor, and a maximum of 2 subsequent chemotherapy treatment. Patients will be screened for baseline anti-β glucan antibody level (ABA; measured in peripheral blood). Those patients with an ABA greater than or equal to 20 mcg/ml and meeting all other I/E criteria, will be enrolled.

The study will enroll 47 patients with 23 patients enrolled into Stage 1. If 4 or more patients in Stage 1 have an objective response after 12 weeks of treatment, the study will proceed into Stage 2. A total of 24 patients will be enrolled in Stage 2 for a total combined population of 47. Overall, objective responses must be observed in 10 patients for the study to be declared a success.

DETAILED DESCRIPTION:
Study PGG-BCA-2121 is a multicenter, open-label, Phase 2 study of patients with metastatic breast cancer who have progressed through prior hormonal therapy with at least one CDK4/6 inhibitor, and a maximum of 2 subsequent chemotherapy treatment. All patients will be immune checkpoint inhibitor-naive.

A total of 47 mBCA patients will be enrolled to treatment with the combination of Imprime PGG 4 mg/kg with pembrolizumab 200mg. Patients will be screened and enrolled if baseline ABA level is greater than or equal to 20 mcg/mL (ABA+) and if all other inclusion/ exclusion criteria are met (ABA is measured in peripheral blood). Approximately 200 patients will be screened (allows for pre/ early screening for ABA levels).

Dosing will occur in three-week cycles. On Day 1 of each cycle, all patients will receive Imprime PGG 4 mg/kg IV over ~ 2-4 hr (based on body weight) followed by pembrolizumab 200 mg, IV over 30 min. On Day 8 and 15 of each cycle, patients will receive only Imprime PGG. Premedications (defined by the protocol) will be administered ~30 min before initiation of Imprime PGG during Cycles 1-3 (thereafter at the physician's discretion). Patients will dose to confirmed progression, safety event, or other administrative reason requiring discontinuation; all patients are allowed to dose up to 35 cycles.

For all patients, a baseline CT/MRI will be conducted. The first scan to assess response will be conducted 12 wks post-initiation of study treatment (pre-Cycle 5) and then q12wks thereafter until confirmed progression or discontinuation. At any time, if a patient's response is progressive disease (PD), the patient will dose for an additional 4-8 wks (physician discretion) followed by a confirmatory scan. If that scan shows progressive disease, the patient will move into overall survival monitoring. Response will be assessed by RECISTv1.1 and iRECIST will be applied by the Investigator solely for clinical management of patients as described below. All scans will be read locally and by blinded central review.

At screening, an official historical diagnostic pathology report +/- archival tissue (formalin-fixed paraffin embedded [FFPE]) will be retrieved to confirm historical diagnosis of ER/PR status. All patients will have a newly obtained core or excisional biopsy at 6 wks after initiation of study treatment. Fresh biopsies at baseline and progression or End of Treatment are strongly encouraged but not mandated. Preferably, biopsies should be non-bone and if amenable, a biopsy of a liver lesion not designated as target or non-target is preferred. Patients with bone only metastases (BOM) are not eligible, except if such lesions have a distinct, associated soft tissue component that is measurable as per RECIST 1.1.

Blood samples for safety monitoring and translational endpoints will be collected on all patients as detailed in the Schedule of Activities.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or legally acceptable representative if applicable) provides written informed consent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have historically confirmed histological diagnosis of metastatic ER/PR+/HER2(-) subtype breast cancer

   1. HR+: Positive for estrogen receptor and/or progesterone receptor staining, indicated by ≥1% immunoreactive tumor nuclei
   2. HER2-: Immunohistochemistry assay demonstrating no or faint staining in ≤10% of tumor cells (IHC score of 0 to 1+) or negative by dual probe in situ hybridization assay
4. Have peripheral blood levels of IgG anti-β-glucan antibody (ABA) of greater than, or equal to 20 mcg/mL as determined by an ELISA test within 90 days prior to start of study treatment.
5. Must have progressed on at least one hormone therapy (AI or SERD) + CDK 4/6 inhibitor (and alpelisib if PIK3CA mutated) and up to two lines of prior chemotherapy (i.e., capecitabine, taxanes). (Patient may have progressed after any number of hormone therapies alone or combined with small molecule inhibitors, i.e., mTOR, PIK3CA, CDK 4/6, etc.)
6. Have documented objective radiographic or clinical disease progression after treatment with estrogen-targeted therapies with at least one CDK4/6 inhibitor.
7. Be willing to provide an archival tissue sample and undergo one on-treatment core or excisional biopsy of a tumor lesion not previously irradiated (Formalin-fixed, paraffin embedded [FFPE]tissue blocks are preferred to slides).
8. Have at least one radiologically measurable lesion as per RECIST v1.1 defined as a lesion that is at least 10 mm in longest diameter imaged by CT scan or MRI and obtained by imaging within 28 days prior to registration. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   a. Note: Patients with bone only metastases (BOM) are not eligible, except if such lesions have a distinct, associated soft tissue component that is measurable as per RECIST 1.1.
9. Have resolution of all previous treatment-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (less than or equal to Grade 2) and alopecia. If the patient received major surgery or radiation therapy of > 30 Gy, must have recovered from the toxicity and/or complications from the intervention.
10. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Have life expectancy of 3 months or greater as determined by the treating physician.
12. Have a negative PCR test at screening for SARS-COV-2 RNA.
13. Have adequate organ function (all screening labs should be performed within 10 days prior to treatment initiation):
14. Female patients of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
15. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies

    1. Not a woman of childbearing potential (WOCBP)
    2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
16. Be willing and have the ability to comply with scheduled visits (including geographical proximity), treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

The patient must be excluded from participating in the trial if the patient:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Has received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks to Study Day 1 (or within 2 weeks for kinase inhibitors or other short half-life drugs), or within 5 half-lives for a prior investigational drug and two weeks from use of an investigational device.

   1. Note: Patients must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Patients with ≤Grade 2 neuropathy may be eligible. Patients with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
   2. Note: If the patient had major surgery, the patient must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention.
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

   c. Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
5. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Note:

   Administration of killed vaccines are allowed.
6. Has had an allogeneic tissue/solid organ transplant.
7. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF, or recombinant erythropoietin) within 4 weeks prior to Study Day 1.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug.
9. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   a. Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
10. Has known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
11. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
12. Had previous exposure to Imprime PGG.
13. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
14. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis/ interstitial lung disease.
15. Has an active infection requiring systemic therapy.
16. Has known history of active tuberculosis.
17. Has a known history of HIV infection. No HIV testing is required unless mandated by local health authority.
18. Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

    a. Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by a local health authority.
19. Has a clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome within ≤ 6 months prior to start of study treatment, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
20. Has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate the patient in the clinical study.
21. Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.
22. A WOCBP who has a positive urine pregnancy test (within 72 hours) prior to treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
23. Is breast feeding or expecting to conceive children within the projected duration of the trial, starting with the prescreening or screening visit through 120 days after the last dose of trial treatment.
24. Is a first-degree relative of the investigator, study staff or study sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Within 24 months of last patient enrolled
  ORR by RECIST v1.1 following treatment with Imprime PGG + pembrolizumab

SECONDARY OUTCOMES:
Median Progression Free Survival (mPFS) | Within 24 months of last patient enrolled
  PFS by RECIST v1.1 following treatment with Imprime PGG + pembrolizumab
PFS at 6, 9, 12, 18, and 24 months | Within 24 months of last patient enrolled
  PFS at 6, 9, 12, 18, and 24 months by RECIST v1.1 following treatment with Imprime PGG + pembrolizumab
Median Overall Survival (mOS) | Within 48 months of last patient enrolled
  Median Overall Survival following treatment with Imprime PGG + pembrolizumab
OS rates at 6, 9, 12, 18, 24 months | Within 24 months of last patient enrolled
  OS rates at 6, 9, 12, 18, 24 months following treatment with Imprime PGG + pembrolizumab
Disease Control Rate (DCR) | Within 24 months of last patient enrolled
  Disease Control Rate by RECIST v1.1 following treatment with Imprime PGG + pembrolizumab
Duration of Response (DoR) | Within 24 months of last patient enrolled
  Duration of Response by RECIST v1.1 following treatment with Imprime PGG + pembrolizumab
Profile safety of Imprime PGG in combination with pembrolizumab | Within 24 months of last patient enrolled
  Safety profile of Imprime PGG in combination with pembrolizumab following treatment with Imprime PGG + pembrolizumab
Correlate changes in immune cell activation markers in tumor samples and in peripheral blood immune cells with treatment outcome | Within 24 months of last patient enrolled
  Correlate phenotypic activation of CD86 (immune cell subsets monocytes, dendritic cells) and T-cell activation (Ki-67, CD38, and HLA-DR) in tumor samples and peripheral blood immune cells with treatment outcome measured by flow cytometry and immunohistochemistry (IHC).
Correlate PD-L1 status and changes in the tumor immune microenvironment with treatment outcome | Within 24 months of last patient enrolled
  Correlate PD-L1 scoring with ORR, OS, and PFS measured by IHC.
Correlate levels of serum anti-β-glucan antibody (ABA) with treatment outcome | Within 24 months of last patient enrolled
  To correlate anti-β-glucan antibody (ABA) concentrations in serum with ORR, OS, and PFS measured by ELISA.
Correlate treatment outcome in select metastatic breast cancer subpopulations | Within 24 months of last patient enrolled
  To correlate treatment outcome with ER/PR positivity (scored from tumor biopsies by IHC at screening and end of cycle 2), prior lines of therapy, and/or comprehensive medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, MD, Study Chair — Stony Brook University
Locations (16):
- United States (16):
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of Colorado at Denver, Denver, Colorado
  - University of Miami and Clinics -Sylvester Comprehensive Cancer Center, Miami, Florida
  - Mt. Sinai (Miami), Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Louisiana State University Health Sciences Center - New Orleans, New Orleans, Louisiana
  - HealthPartners Cancer Research Center, Saint Louis Park, Minnesota
  - St. Luke's Cancer Institute, Kansas City, Missouri
  - St. Vincent - Frontier Cancer Center, Billings, Montana
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Columba University Medical Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Thomas Jefferson University- Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No